CLINICAL TRIAL: NCT06162312
Title: Efficacy of Antenatal Perineal Massage in Reducing Postpartum Morbidities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 182/2566
Record Dates: First submitted 2023-12-01; First posted 2023-12-08 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2023-12

CONDITIONS: Perineum; Injury; Anal Incontinence; Urinary Incontinence
Keywords: antenatal perineal massage; postpartum morbidities; Anal Incontinence
MeSH Terms: conditions — Wounds and Injuries; Encopresis; Urinary Incontinence

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antenatal perineal massage (Experimental): daily 5-minute perineal massage from the 34th or 35th week of pregnancy until delivery
  Interventions: Other: Antenatal perineal massage
- Control (No Intervention): standard antenatal, intrapartum and postpartum care

INTERVENTIONS:
Other: Antenatal perineal massage — Participants at 34-35 weeks of gestation were received training in self-perineal massage and performed a daily 5-minute massage using water-based jelly until delivery to compare with standard obstetric care on postpartum morbidities
  Arms: Antenatal perineal massage

SUMMARY:
A randomized controlled trial was undertaken at Rajavithi Hospital, Bangkok, Thailand, encompassing 106 primigravidae within the period of December 2023 to June 2024. The intervention group underwent antepartum perineal massage, starting at the 34th - 35th week of gestation and extending until delivery, while the control group did not receive such intervention. The primary outcome evaluated was the incidence of anal incontinence at the 3-month postpartum. Secondary outcomes included the duration of each labor stage, perineal tears and their degrees, episiotomy occurrences, Apgar scores at 1 and 5 minutes, postpartum pain within 24 hours, dyspareunia, and urinary incontinence at the 3-month postpartum.

DETAILED DESCRIPTION:
Vaginal births often result in perineal trauma, leading to substantial morbidity. This study hypothesized that antenatal perineal massage (APM) could mitigate the incidence of perineal injuries and related postpartum morbidities.

Participants at 34-35 weeks of gestation were randomly assigned by a computer program to either the Antenatal Perineal Massage (APM ) group or the control group. The APM group received training in self-perineal massage and performed a daily 5-minute massage using water-based jelly until delivery, while the control group did not receive such intervention.

The technique involved inserting the thumb finger 3-5 cm into the vagina, using a water-based jelly for lubrication. The procedure included maintaining the thumb steady on the perineum for 1 minute, applying up-and-down pressure for 1 minute, and performing downward and sideways sweeping motions for 3 minutes. Initial massage sessions were conducted under supervision at the antenatal clinic.

Participants were advised to discontinue APM in case of premature rupture of membranes (PROM), bleeding, or infection, seeking prompt hospital management. Additionally, they were instructed to maintain a diary documenting their daily APM sessions.

Both groups received standard antenatal, intrapartum, and postpartum care. Obstetric care providers, investigator and outcomes assessor remained blinded to participants' study group allocations.

During labor at the casualty department, routine care was administered without intervention in labor management or cesarean delivery decisions. Recorded data encompassed the duration of each labor stage, perineal tears and their degrees, episiotomy occurrences, urgency for cesarean section or operative vaginal delivery, infant weight, sex, Apgar scores at 1 and 5 minutes, and postpartum pain using a verbal numerical rating scale within 24 hours.

Participants were followed up at 3 months post-delivery to evaluate the anal incontinence, urinary incontinence (assessed via the validated Thai version of Pelvic Floor Distress Inventory - 20 (PFDI-20)), and dyspareunia (using a verbal numerical rating scale

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous singleton pregnant women older than 18 years at 34 - 35 weeks of gestation
* The fetus has a cephalic presentation.
* Proficiency in the Thai language for communication
* Willingness to engage in research projects
* Intending to deliver at Rajavithi Hospital

Exclusion Criteria:

* Genital infections such as herpes or candida vulvovaginitis.
* Previous Caesarean section.
* Pregnant women who underwent epidural anesthesia or required instrumental delivery
* Pregnant women with a history of chronic cough, urinary incontinence, Anal incontinence, pelvic floor dysfunction, or connective tissue diseases
* Contraindications to vaginal childbirth, such as placenta previa or Placenta accreta spectrum disorder
* Birth before arrival

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Anal incontinence | At 3 months post-delivery
  To compare anal incontinence between intervention group and control group. Assessed via the validated Thai version of Pelvic Floor Distress Inventory - 20 (PFDI-20)

SECONDARY OUTCOMES:
Urinary incontinence | At 3 months post-delivery
  To compare urinary incontinence between intervention group and control group. Assessed via the validated Thai version of Pelvic Floor Distress Inventory - 20 (PFDI-20)
Dyspareunia | At 3 months post-delivery
  To compare dyspareunia between intervention group and control group. Assessed via the verbal numerical rating scale
Postpartum pain | At 24 hours post-delivery
  To compare postpartum pain between intervention group and control group. Assessed via the verbal numerical rating scale
Duration of each labor stage | During delivery
  To compare duration of first, second and third stage of labor stage between intervention group and control group.
Perineal tears and their degrees | During delivery
  To compare perineal tear occurrences and their degrees between intervention group and control group.
Episiotomy | During delivery
  To compare episiotomy occurrences between intervention group and control group.
Apgar scores | During delivery
  To compare Apgar scores at 1 and 5 minutes of the newborns between intervention group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi hospital, Phaya Thai, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ugwu EO, Iferikigwe ES, Obi SN, Eleje GU, Ozumba BC. Effectiveness of antenatal perineal massage in reducing perineal trauma and post-partum morbidities: A randomized controlled trial. J Obstet Gynaecol Res. 2018 Jul;44(7):1252-1258. doi: 10.1111/jog.13640. Epub 2018 Apr 2. PMID 29607580
- [Background] Bunyavejchevin S, Ruanphoo P. Thai translation and validation of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) and Pelvic Floor Distress Inventory (PFDI-20). Int Urogynecol J. 2022 Nov;33(11):3137-3142. doi: 10.1007/s00192-022-05148-y. Epub 2022 Apr 7. PMID 35389055
- [Background] Steiger A, Rupprecht R, Spengler D, Guldner J, Hemmeter U, Rothe B, Damm K, Holsboer F. Functional properties of deoxycorticosterone and spironolactone: molecular characterization and effects on sleep-endocrine activity. J Psychiatr Res. 1993 Jul-Sep;27(3):275-84. doi: 10.1016/0022-3956(93)90038-4. PMID 8295159
- [Background] Nadkarni TD, Goel A, Shenoy A, Karapurkar AP. Cladosporium bantianum (trichoides) infection of the brain. J Postgrad Med. 1993 Jan-Mar;39(1):43-4. PMID 8295150
- [Background] Tom BH, Macek CM, Subramanian C, Miller AL, Sengupta J. In vitro expression of suppressogenic and enhancing activities in human colon cancer cells. J Biol Response Mod. 1984 Aug;3(4):435-44. PMID 6481402
- [Background] Dieb AS, Shoab AY, Nabil H, Gabr A, Abdallah AA, Shaban MM, Attia AH. Perineal massage and training reduce perineal trauma in pregnant women older than 35 years: a randomized controlled trial. Int Urogynecol J. 2020 Mar;31(3):613-619. doi: 10.1007/s00192-019-03937-6. Epub 2019 Apr 2. PMID 30941442
- [Background] Mei-dan E, Walfisch A, Raz I, Levy A, Hallak M. Perineal massage during pregnancy: a prospective controlled trial. Isr Med Assoc J. 2008 Jul;10(7):499-502. PMID 18751626
- [Background] Abdelhakim AM, Eldesouky E, Elmagd IA, Mohammed A, Farag EA, Mohammed AE, Hamam KM, Hussein AS, Ali AS, Keshta NHA, Hamza M, Samy A, Abdel-Latif AA. Antenatal perineal massage benefits in reducing perineal trauma and postpartum morbidities: a systematic review and meta-analysis of randomized controlled trials. Int Urogynecol J. 2020 Sep;31(9):1735-1745. doi: 10.1007/s00192-020-04302-8. Epub 2020 May 12. PMID 32399905
- [Background] Tin RY, Schulz J, Gunn B, Flood C, Rosychuk RJ. The prevalence of anal incontinence in post-partum women following obstetrical anal sphincter injury. Int Urogynecol J. 2010 Aug;21(8):927-32. doi: 10.1007/s00192-010-1134-0. Epub 2010 Apr 27. PMID 20422153